CLINICAL TRIAL: NCT04335773
Title: COVID-19 in Hospitalised Norwegian Children - Risk Factors, Outcomes and Immunology
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Collaborators: St. Olavs Hospital (Other); Helse Stavanger HF (Other Government); Haukeland University Hospital (Other); University Hospital of North Norway (Other); Alesund Hospital (Other); Norwegian Institute of Public Health (Other Government); The University of New South Wales (Other); University of Bristol (Other); Sykehuset Ostfold (Other); Nordlandssykehuset HF (Other); Vestre Viken Hospital Trust (Other); Helse Fonna (Other); Helse Nord-Trøndelag HF (Other); Oslo University Hospital (Other); Sykehuset Innlandet HF (Other)
Responsible Party: Principal Investigator, Christopher Inchley, Principal investigator, University Hospital, Akershus
Other Study IDs: 20/03794
Record Dates: First submitted 2020-04-03; First posted 2020-04-06 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Pediatric Respiratory Diseases; COVID; Fatigue Post Viral

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Blodsamples, Eluate from nasopharyngeal sample, Urin, Feces,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sars-CoV-2 positive: Children positive for SARS-CoV-2
- SARS-CoV-2 negative: Children negative SARS-CoV-2

SUMMARY:
Prospective cohort study of COVID-19 infection among children in Norway.

DETAILED DESCRIPTION:
This nation-wide, prospective cohort study of COVID-19 infection addresses three main issues: 1) Epidemiological risk factors; 2) Natural history (including immunological mechanisms and long term effects) and 3) Support of infection prevention. Also, the study focuses solely on children.

Children (0-18 years of age) admitted to hospital with suspected COVID-19 are eligible (Fig. 1). Those with confirmed COVID-19 serve as cases, whereas those with non-COVID-19 serve as controls; both groups will be followed prospectively for 6 months. Three objectives/Work Packages (WPs) are defined:

* In WP1, the investigators will investigate risk factors for severe outcome of the acute infection; potential risk factors include sex, age, comorbidities, initial clinical findings, infectious load, and genetic markers.
* In WP2, the investigators will investigate the immunological response to acute infection, focusing on initial innate host response and its associations to inflammatory enhancement, genetic factors and clinical course.
* In WP3, the investigators will investigate the prevalence and risk factors of long-lasting complication, in particular the development of post-infectious chronic fatigue

ELIGIBILITY:
Inclusion Criteria:

Suspected covid-19 infection and age 0-18 years

Exclusion Criteria:

Age >18 years

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children seeking hospital care i Norway
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2020-04-03 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Risk Factors for severe infection | 2030
  Identify comorbidities predisposing for severe infection
Immunulogical mechanisms | 2030
  Immunological response to acute infection, focusing on initial innate host response and its associations to inflammatory enhancement, genetic factors and clinical course.
Long term outcome | 2030
  prevalence and risk factors of long-lasting complication, in particular the development of post-infectious chronic fatigue

CONTACTS AND LOCATIONS:
Locations (1):
- Akershus universistetssykehus, Lørenskog, Norway